CLINICAL TRIAL: NCT05592210
Title: Influence and Mechanism of Dyadic Coping on Parenting Stress and Parenting Self-Efficacy in Parents of Preterm Infant
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Wei XIA, PhD, Associate professor, Sun Yat-sen University
Other Study IDs: preterm infant（PES）
Record Dates: First submitted 2022-10-20; First posted 2022-10-24 (Actual); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Premature Infant Disease
Keywords: Premature Infant; Parental self-efficacy; Parenting Stress; Dyadic Coping
MeSH Terms: conditions — Premature Birth | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Questionnaires assessed Parents of preterm infants: Inclusion criteria for parents
  1. Parents of hospitalized preterm infants with a gestational age of less than 37 weeks;
  2. Both parents are at least 18 years old;
  3. Able to read and communicate in Chinese, able to complete the questionnaire independently or with the help of the investigator;
  Inclusion criteria for infant
  1. Gestational age less than 37 weeks;
  2. admitted to the NU or NICU and discharged after treatment;
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — Participants will be asked to fill out the the Demographic Information Sheet, Karitane parenting confidence scale, Parental Stressor Scale: Neonatal Intensive Care Unit (PSS:NICU) and Dyadic Coping Inventory.

SUMMARY:
The goal of this observational study is to investigate the parenting stress, parenting self-efficacy and dyadic coping of preterm parents and explore the influence and pathway analysis of dyadic coping between parenting stress and parenting self-efficacy.

DETAILED DESCRIPTION:
For now, there is a lack of investigation and research on parenting stress, parenting self-efficacy and dyadic coping of co-parenting for discharged premature infants in the literature, and the mediating effect of dyadic coping between parenting stress and parenting self-efficacy of preterm parents has not been verified yet. This study aims to provide a theoretical basis for effective intervention for preterm parents with high parenting pressure and insufficient parenting self-efficacy in clinical work.

ELIGIBILITY:
Inclusion criteria for parents

* Parents of hospitalized preterm infants with a gestational age of less than 37 weeks;
* Both parents are at least 18 years old;
* Able to read and communicate in Chinese, able to complete the questionnaire independently or with the help of the investigator;

Inclusion criteria for Infants

* Gestational age less than 37 weeks;
* admitted to the NU or NICU and discharged after treatment

Exclusion criteria for parents

* Single-parent family;
* Parents diagnosed with severe anxiety and depression;

Exclusion criteria for Infants

* for birth defects cannot be cured and affect the quality of life;
* infants who were given up treatment due to illness or family reasons;
* transferred or death;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The parents of premature infants admitted to Peking University Shenzhen Hospital from November 2022 to November 2023.
Sampling Method: Non-Probability Sample
Enrollment: 308 (Estimated)
Dates: Start 2023-03-16 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Karitane parenting confidence scale | baseline
  The Karitane parenting confidence scale will measure the Parenting Self-efficacy of preterm parents. The scale adopts a Likert 4-level scoring method, with 0 representing hardly ever and 3 representing most of the time. The higher the scores of each dimension and the total score, the higher the self-efficacy of the Parenting Self-efficacy of preterm parents.
Parental Stressor Scale: Neonatal Intensive Care Unit (PSS:NICU) | baseline
  The Parenting Stress of preterm parents will be measured by Parental Stressor Scale: Neonatal Intensive Care Unit (PSS: NICU). The scale was scored from 1(not experient) to 5(extremely stressful) points, and the higher the score, the higher the feeling of parenting stress.
Dyadic Coping Inventory | baseline
  The Dyadic Coping of preterm parents will be measured by Dyadic Coping Inventory. The total score ranges from 36 to 180.. The higher the score, the more supportive behaviors the partner gives.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xia, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Peking University Shenzhen Hosipital, Shenzhen, China

IPD SHARING:
Plan to Share IPD: No